CLINICAL TRIAL: NCT04278469
Title: A Prospective, Randomized, Comparative Study to Evaluate Efficacy of Anticancer Chemotherapy in Predicting Prognosis and Determining Chemotherapy Method in Early Hormone Receptor-positive Breast Cancer Patients With Clinicopathological High Risk and GenesWell™ BCT Low Risk at Multi-center in Korea
Brief Title: Clinical High and Genomic Low Hormone Receptor-positive Early Breast Cancer Patients With or Without Adjuvant Chemotherapy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Gencurix, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GCX-BCT-06
Record Dates: First submitted 2020-02-18; First posted 2020-02-20 (Actual); Last update posted 2020-02-20 (Actual); Status verified 2020-02

CONDITIONS: Early Hormone Receptor-positive Breast Cancer
MeSH Terms: interventions — Antineoplastic Agents

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients with chemotherapy (Active Comparator)
  Interventions: Drug: Chemotherapy Drugs, Cancer
- Patients without chemotherapy (No Intervention)

INTERVENTIONS:
Drug: Chemotherapy Drugs, Cancer — Clinical high and genomic low Hormone Receptor-positive early breast cancer patients with or without adjuvant chemotherapy
  Other Names: GenesWell™ BCT (analysis genomic risk)
  Arms: Patients with chemotherapy

SUMMARY:
A prospective, randomized, comparative study to evaluate efficacy of anticancer chemotherapy in predicting prognosis and determining chemotherapy method in early Hormone Receptor-positive breast cancer patients with clinicopathological high risk and GenesWell™ BCT low risk at multi-center in Korea

ELIGIBILITY:
Inclusion Criteria:

1. Adult women aged 19-80 at screening
2. Histologically invasive carcinoma
3. Hormone receptor positive (Estrogen, ER+ and/or Progesterone, PR+)
4. Human epidermal growth factor receptor 2 negative (HER2-)
5. Axillary lymph node assessment: pN0 or pN1
6. Tumor size≥0.5cm
7. Clinical high risk (based on modified Adjuvant! Online)
8. Patients who agree to genetic testing
9. Patients who have adequate organ function
10. Genomic low risk (based on GenesWell BCT)
11. De novo primary cancer
12. Patients how performed surgery with curative aim
13. Patients who have provided written informed consent themselves

Exclusion Criteria:

1. Hormone receptor negative (Estrogen, ER- and Progesterone, PR-)
2. Human epidermal growth factor receptor 2 positive (HER2+)
3. Axillary lymph node assessment: pN2 or pN3
4. Patients who are received chemotherapy prior to operation
5. Patients who are received radiotherapy prior to operation
6. Tumor size<0.5cm
7. Clinical low risk
8. FFPE tumor sample is not available
9. Patients with following conditions:

   * Patient with chronic liver disease
   * Patient with cerebrovascular disease
   * Patient with chronic mental disorder
   * Pregnant women, women of childbearing potential or lactating women
10. Patients who are deemed inappropriate as study participants by investigators
11. Patients with recurrent breast cancer or treatment history of breast cancer
12. Patients who have not undergone surgery

Ages: 19 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 194 (Estimated)
Dates: Start 2019-01-11 (Actual); Primary Completion 2029-01 (Estimated); Study Completion 2029-01 (Estimated)

PRIMARY OUTCOMES:
10-year distant metastasis free survival | up to 10 years
  To evaluate 10-year distant metastasis free survivals according to adjuvant chemotherapy in patients with clinical high and genomic low risk

SECONDARY OUTCOMES:
disease free survival | up to 10 years
  To evaluate 10-year disease free survivals and overall survivals according to adjuvant chemotherapy in patients with clinical high and genomic low risk
overall survival | up to 10 years
  To evaluate 10-year disease free survivals and overall survivals according to adjuvant chemotherapy in patients with clinical high and genomic low risk

CONTACTS AND LOCATIONS:
Locations (1):
- Samsung Medical Center, Seoul, South Korea